CLINICAL TRIAL: NCT00404937
Title: Tobradex BID Compared to TOBRADEX and TOBREX/Vehicle
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-05-60
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2007-09

CONDITIONS: Post-surgical Inflammation
MeSH Terms: interventions — Tobramycin, Dexamethasone Drug Combination

INTERVENTIONS:
Drug: Tobradex (Antibiotic steroid combination)

SUMMARY:
The purpose of this study is to compare the new formulation of Tobradex to the current approved formulation

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cataract extraction

Exclusion Criteria:

* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Anterior chamber inflammation

SECONDARY OUTCOMES:
Aqueous cells and flare
ocular pain
physician's impression of infection
frequency of treatment failures